CLINICAL TRIAL: NCT05719051
Title: Effect of Albumin Infusion in Patients With Decompensated Cirrhosis Hospitalized for Treatment of Complications of Liver Disease
Brief Title: Albumin Infusion in Inpatients With Decompensated Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Qing XIe, Professor, Ruijin Hospital
Other Study IDs: RJH-Albumin
Record Dates: First submitted 2023-01-08; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Decompensated Cirrhosis; Acute-On-Chronic Liver Failure
Keywords: Albumin; decompensated cirrhosis; Systemic inflammation; Prognosis
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- High-dose group: Total Intravenous albumin infusion >1.5g/kg per week while hospitalization
  Interventions: Drug: Albumin infusion
- Medium-dose group: Total Intravenous albumin infusion 1.0 to 1.5g/kg per week while hospitalization
  Interventions: Drug: Albumin infusion
- Low-dose group: Total Intravenous albumin infusion <1.0g/kg per week while hospitalization
  Interventions: Drug: Albumin infusion

INTERVENTIONS:
Drug: Albumin infusion — Albumin infusion was administrated according to the standard clinical practice

SUMMARY:
Albumin infusion in patients with hospitalized decompensated, even in short-term period use, could improve survival through the reduction of systemic inflammation, which is the main driver of acute-on-chronic liver failure in cirrhosis. The effects could be highly associated with the albumin dosage. A comprehensive evaluation of the inflammation response by robust measurement is needed to prove insights into the therapeutic implications of albumin infusion.

The purpose of this study is to compare the effects of different amount of human albumin infusion per week in patients with hospitalized decompensated cirrhosis on 28-day transplant-free survival and to further compare the alleviation of inflammation, reduction of incidence of nosocomial infection, spontaneous bacterial peritonitis (SBP), acute kidney injury (AKI), acute-on-chronic liver failure (ACLF), and 90-day transplant-free survival. This will be a multicenter, national, retrospective study. There will be no randomization in this retrospective study. All patients who meet the inclusion criteria and not the exclusion criteria will be enrolled. All identified patients who meet criteria will be given an ID number comprised of a site number and patient number.

DETAILED DESCRIPTION:
Patients with decompensated cirrhosis frequently develop various complications, be it related to salt and water retention, renal dysfunction, hepatic encephalopathy, portal hypertensive bleeds, or various infections. These lead to frequent hospital admissions, impaired quality of life, and increased morbidities and mortality.

Although recent investigations have helped to elucidate the pathogenetic mechanisms that lead to the development of these complications, exactly how much each of these pathogenetic mechanisms contributes to the development of these complications is not clear. Among them, hypoalbuminemia has long been considered a cardinal feature of decompensated cirrhosis.

Human albumin is the main modulator of fluid distribution among the body compartments and also exerts many other biological properties unrelated to its oncotic power including antioxidation, immune modulation and anti-inflammatory effect, and endothelial stabilization as well as vascular integrity. Albumin infusion has been recommended by international guidelines after large-volume paracentesis in patients with ascites, or in spontaneous bacterial peritonitis to prevent and treat the hepatorenal syndrome. Long-term prophylactic administration of albumin to outpatients with prior history of ascites is also effective in preventing further complications and improving survival. A subsequent study suggests an anti-inflammatory effect of albumin in patients with cirrhosis; this finding suggests that infusions of albumin might increase survival by limiting systemic inflammation.

These promising data suggested a disease-modifying agent role of albumin in patients with decompensated cirrhosis. The investigators, therefore, hypothesized that albumin infusion in patients with hospitalized decompensated, even in short-term period use, could also improve survival through the reduction of systemic inflammation, which is the main driver of acute-on-chronic liver failure in cirrhosis. The effects could be highly associated with the albumin dosage. A comprehensive evaluation of the inflammation response by robust measurement is needed to prove insights into the therapeutic implications of albumin infusion.

To test these hypotheses, the investigators planned to perform retrospective analysis in two established cohorts of hospitalized decompensated cirrhosis: 1) the "RJH" cohort of decompensated cirrhosis in Ruijin Hospital enrolled between 2016 and 2018; 2) an established cohort of inpatients with cirrhosis enrolled from 23 centers in China between 2018 and 2019 (the "SONIC" study).

ELIGIBILITY:
Inclusion Criteria:

Patients with decompensated cirrhosis nonelective admitted for overt ascites, active gastrointestinal bleeding, hepatic encephalopathy, bacterial/fungal infection, or jaundice, etc.

Exclusion Criteria:

1. Age below 16 or over 80 years
2. Lactation/ Pregnancy women
3. HIV infection
4. Admitted for scheduled procedures (e.g., band ligation, splenectomy, transjugular intrahepatic portosystemic shunting, liver biopsy) or reexamination or multidisciplinary consultation)
5. Hepatocellular carcinoma (HCC) outside Milan criteria or other disseminated malignancies
6. Previous liver transplantation
7. With previously known severe extra-hepatic diseases (e.g., chronic renal failure requiring hemodialysis, severe heart disease; severe chronic pulmonary disease, psychiatric disorders)
8. Taking immunosuppressive or anticoagulation drugs for the treatment of extra-hepatic disease.
9. Patient' s refusal to participation
10. Failure to provide prior informed consent or with documented evidence that the patient has no legal surrogate decision maker and it appears unlikely that the patient will regain consciousness or sufficient ability to provide delayed informed consent

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Based on the ID card
Study Population: Target population is hospitalized patients with decompensated cirrhosis. For the purpose of this study, two established prospect cohorts will be used retrospectively including the "RJH" cohort and the "SONIC" cohort. All patients in the abovementioned cohorts had at least one of the following events for inclusion: overt ascites, active gastrointestinal bleeding, hepatic encephalopathy, bacterial/fungal infection, or jaundice.
Sampling Method: Probability Sample
Enrollment: 564 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Transplant-free survival at day 28 since enrollment | From enrollment (Day 1) to Day-28
  Transplant-free survival at day 28 since enrollment

SECONDARY OUTCOMES:
Changes of inflammatory markers from baseline | From baseline (sample collection date) to Day 7 and Day 14, respectively
  Changes of the level of each measured inflammatory marker (IL6, IL-8, TNF-a, etc.) at Day 7 and Day 14 as compared to the baseline level.
Cumulative incidence of nosocomial infection by day 28 | From enrollment (Day 1) to Day-28
  Cumulative incidence of nosocomial infection by day 28
Cumulative incidence of SBP by day 28 | From enrollment (Day 1) to Day-28
  Cumulative incidence of SBP by day 28
Cumulative incidence of AKI by day 28 | From enrollment (Day 1) to Day-28
  Cumulative incidence of AKI by day 28
Cumulative incidence of ACLF by day 28 | From enrollment (Day 1) to Day-28
  Cumulative incidence of ACLF by day 28
Transplant-free survival at day 90 since enrollment | From enrollment (Day 1) to Day-90
  Transplant-free survival at day 90 since enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Diseases , Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No